CLINICAL TRIAL: NCT03234686
Title: Deferiprone to Delay Dementia (The 3D Study): a Clinical Proof of Concept Study
Brief Title: Deferiprone to Delay Dementia (The 3D Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neuroscience Trials Australia (Other)
Collaborators: The Florey Institute of Neuroscience and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DEF001
Record Dates: First submitted 2017-07-23; First posted 2017-07-31 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Mild Cognitive Impairment; Prodromal Alzheimer's Disease; Mild Alzheimer's Disease
Keywords: Dementia; Alzheimer's Disease
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Alzheimer Disease | interventions — Deferiprone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deferiprone (Experimental): Patients will orally receive the equivalent 15 mg/kg of 600mg delayed release Deferiprone tablets twice daily.
  Interventions: Drug: Deferiprone 600mg delayed release tablets
- Placebo (Placebo Comparator): Patients will receive matching placebo tablets designed to mimic the experimental treatment, twice daily
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Deferiprone 600mg delayed release tablets — The active substance, Deferiprone, is a member of the 3-hydroxypyrid-4-one class of iron chelators, which have a high affinity for ferric iron, binding it in a 3:1 (Deferiprone:iron) molar ratio.
  Arms: Deferiprone
Drug: Placebo Oral Tablet — The placebo will mimic the Deferiprone arm in every way, except the placebo will not include the active ingredient
  Arms: Placebo

SUMMARY:
This study is a phase 2, randomised, placebo-controlled, multicentre study to investigate the safety and efficacy of Deferiprone in participants with Prodromal Alzheimer's Disease (pAD) and Mild Alzheimer's Disease (mAD). In this phase 2 study, the investigators aim to determine whether Deferiprone (15 mg/kg BID orally) slows cognitive decline in Alzheimer's patients. As secondary outcomes, safety and iron levels in the brain will be evaluated.

DETAILED DESCRIPTION:
This Phase II study is designed as a randomised, double-blinded, placebo controlled, multi-centre study for subjects with evidence of amyloid positive pAD or mAD.

Participants will be assigned randomly to two groups (Group 1 Deferiprone (15mg/kg BID orally), Group 2: Placebo). Participants will have a 2 in 3 chance to be placed in the Deferiprone group.

The study will enrol approximately 171 participants over 4 sites in Australia. The overall duration for patients will be 54 weeks. This includes a 55-day screening period, and visits on Day 1, weeks 13, 26, 38,52, and a two-week follow-up visit.

Participants will be screened for the study after signing the approved informed consent form. As part of the 55-day screening phase, subjects will undertake an extensive medical and neurological assessments as well as a PET scan.

At the baseline visit, following the screening phase, blood and urine will be taken for safety monitoring and for measuring APOE-4 gene status. Baseline signs and symptoms will be collected. An MRI will be performed All patients will start with study medication at the Baseline visit.

Participants will return to the centre on Weeks 13, 26, 38, 52 (or early termination) to undertake a neurological examination as well as an assessment of blood samples taken at the visit.

Participants must also attend weekly blood tests.

SAE's, AE's and changes to concomitant medications will be observed and evaluated throughout the study. Each study visit will have a 7-day window after the due date to account for scheduling conflicts/holidays/weekends.

Participants will be given additional study product to account for the 7-day window.

Participants must attend the weekly pathology visits with a 3-day window of the scheduled date or risk termination from the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent in accordance with federal, local and institutional guidelines. For subjects unable to provide written consent, consent will be provided by the Person Responsible per local regulations.
2. Age ≥65 years, or ≥55 years if they have been diagnosed by a psychiatrist or neurologist with dementia, or if they have a validated previous positive amyloid PET scan.
3. Weight between 40 and 120 kg
4. Have an available caregiver
5. Have ≥ 6 years of education (any) and able to follow testing instructions.
6. Have visual and auditory acuity sufficient to perform neuropsychological testing.
7. Have prior evidence of AD pathology, by a positive amyloid assessment, or amyloid PET scan.
8. Demonstrate abnormal memory function in the last 6 months or at screening: International Shopping List Test (ISLT) >1.5 SD below the age adjusted mean
9. Subjective or clinical history of retrospective cognitive decline ≥6 months
10. Evidence of mild symptomatology, as defined by a screening MMSE score of ≥ 20 points
11. Meet National Institute on Ageing/Alzheimer's Association Diagnostic Guidelines for Alzheimer's Disease (NIAAA) research criteria for mAD or pAD
12. If receiving medication for symptomatic AD, have a stable dosing regimen for 3 months prior to screening.
13. Females of Child Bearing Potential (FCBP) must have confirmed negative serum pregnancy test within the 21 days prior to randomization.
14. FCBP and male subjects who are sexually active with FCBP must agree to use highly effective contraception during the study and until 90 days after the last dose of treatment (for sexually active male participants whose partners are FCBP) or until 30 days after the last dose of treatment (for women of childbearing potential participants).

Exclusion Criteria:

1. Clinically significant haematological disorder, including moderate or severe anaemia (blood haemoglobin <110 g/L, WHO definition)
2. Iron deficiency (serum ferritin < 10 ng/mL)
3. Clinically significant abnormal haematological results (sufficiently outside the normal range to warrant further investigation). Mild anaemia (haemoglobin ≥110 g/L) is not an exclusion.
4. Clinically significant abnormal renal or liver function results (sufficiently outside the normal range to warrant further investigation)
5. Presence of non-AD condition that may affect cognition, such as but not limited to Parkinson's Disease (PD), normal pressure hydrocephalus, sleep apnoea requiring O2 treatment
6. Clinically evident vascular disease that could potentially affect the brain, such as but not limited to significant carotid or vertebral stenosis, aortic aneurysm, cerebral haemorrhage
7. History of any stroke in the past 2 years, or transient ischemic attack within the last 6 months
8. History of persistent neurologic deficit, intracranial tumour or structural brain damage
9. History of infection that could affect brain function (eg HIV and syphilis)
10. Autoimmune disorders that potentially cause progressive neurologic disease with associated cognitive deficits, such as but not limited to multiple sclerosis, lupus
11. Major psychiatric illness (depression is acceptable if patient has not had an episode within the past year or is considered in remission or controlled by treatment)
12. A history of relapsing neutropenia.
13. Presence of agranulocytosis or with a history of agranulocytosis
14. Known hypersensitivity to DFP or excipients.
15. Alcohol and/or substance abuse
16. MRI evidence of clinically-significant cerebrovascular pathology. Focal white matter lesions, ≤ 2 lacunar infarcts in non-critical sites and other minor pathology assessed by the investigator to not be causing the current cognitive impairment, will not lead to exclusion.
17. Active major medical illness
18. FCBP not using adequate method of contraception or who is pregnant or nursing
19. Inability to provide informed consent
20. Participation in another clinical trial within 3 months prior to inclusion in the study
21. Subjects for whom MRI is contraindicated (severe claustrophobia, pacemaker, incompatible surgical material, unmovable electronic pump implant)
22. Negative amyloid PET scan or CSF in the last 2 years.
23. Hospital Anxiety and Depression Scale (scores > 8/21 are disqualified).
24. Subject cannot commit to regular blood tests with the interval between tests not exceeding 10 days from the scheduled visit for the duration of the study.
25. Subject has planned surgery which does not permit regular blood tests with the interval between tests not exceeding 10 days from the scheduled visit.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 81 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Efficacy of Deferiprone | 12 months
  Comparison of the efficacy of Deferiprone (15 mg/kg) administered orally twice a day with a matching placebo in subjects with pAD (MCI with brain amyloid pathology) or mAD at 12 months relative to baseline. This will be measured by a series of paper and electronic assessments called the NTB

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | 12 months
  Safety and tolerability will be assessed by the incidence and severity of AEs and changes from baseline of all relevant parameters, including clinical laboratory values, vital signs, ECG and other safety biomarkers. Severity of AEs will be assessed according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 4.03. All subjects will be monitored for AEs until resolution.
Brain Iron Levels | 12 months
  Using MRI to compare iron levels in various brain regions of the Deferiprone and placebo treatment groups at baseline and 12 months.

OTHER OUTCOMES:
The effect of Deferiprone on the episodic memory, executive function and attention composites | 12 months
  Measured by scores on the NTB at 12 months relative to baseline
The Association with Iron levels in the Brain and Cognitive Decline | 12 months
  Using MRI to evaluate if cognitive performance is associated with a change in iron levels over a 12-month period relative to baseline.
The Potential for Brain Iron Load to be Used to Stratify Responsiveness to Deferiprone | 12 months
  Measured by baseline iron MRI and change in cognitive ability from baseline at 12 months.
The Potential for APOE Genotype to be Used to Stratify Responsiveness to Deferiprone | 12 months
  Measured by APOE genotype and changes in cognitive ability from baseline at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ashley I. Bush, Principal Investigator — The Florey Institute of Neuroscience and Mental Health
Locations (8):
- Australia (8):
  - KaRa Institute of Neurological Diseases, Macquarie Park, New South Wales
  - Hunter New England Local Health District, Waratah, New South Wales
  - Box Hill Hospital, Box Hill, Victoria
  - Austin Health, Heidelberg, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - NeuroCentrix, Noble Park, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Australian Alzheimer's Research Foundation, Nedlands, Western Australia

REFERENCES:
- [Derived] Ayton S, Barton D, Brew B, Brodtmann A, Clarnette R, Desmond P, Devos D, Ellis KA, Fazlollahi A, Fradette C, Goh AMY, Kalinowski P, Kyndt C, Lai R, Lim YY, Maruff P, O'Brien TJ, Rowe C, Salvado O, Schofield PW, Spino M, Tricta F, Wagen A, Williams R, Woodward M, Bush AI. Deferiprone in Alzheimer Disease: A Randomized Clinical Trial. JAMA Neurol. 2025 Jan 1;82(1):11-18. doi: 10.1001/jamaneurol.2024.3733. PMID 39495531